CLINICAL TRIAL: NCT06618053
Title: The Cost-effectiveness of Stapes Surgery for Otosclerosis Performed Under Local Versus General Anesthesia
Acronym: CESSO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/879
Record Dates: First submitted 2024-06-10; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Otosclerosis
MeSH Terms: conditions — Otosclerosis | interventions — Cost-Effectiveness Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stapes surgery performed under local anesthesia
  Interventions: Other: cost-effectiveness and audiometry outcomes
- stapes surgery performed under general anesthesia
  Interventions: Other: cost-effectiveness and audiometry outcomes

INTERVENTIONS:
Other: cost-effectiveness and audiometry outcomes — Evaluate cost-effectiveness of stapes surgery performed under local anesthesia as well as evaluate audiometry outcomes

SUMMARY:
Otosclerosis is a localized disorder of the otic capsule, characterized by bone resorption anterior to the oval window in the region of the fissula ante fenestram. This process leads to new sclerotic bone formation, resulting in stapes footplate fixation. It is one of the most common causes of progressive conductive hearing loss in young adults between the age of 30 and 50 year-old. As the disease advances, hearing loss can become mixed and even purely sensorineural due to the pathological process extending into the cochlea.

Stapes surgery is the gold standard procedure for restoring mechanical sound transmission through the middle ear. For patients who are not candidates for surgery, hearing aids offer a valid alternative. Over the years, stapes surgery has evolved into a minimally invasive procedure that can be safely performed as day surgery, under either local or general anesthesia.

The COVID-19 crisis has exacerbated a shortage in anesthesiology teams, limiting operating room availability. To address this issue, stapes surgery for otosclerosis under local anesthesia were increasingly performed. Local anesthesia has several advantages: it allows for immediate hearing tests after prosthesis placement, enabling early detection and correction of vertigo caused by prosthesis displacement, thus minimizing major complications. Additionally, local anesthesia reduces exposure to general anesthesia, thereby decreasing postoperative morbidities.

While there are few studies comparing outcomes and complications of stapes surgery based on the type of anesthesia, a systematic review in 2013 found no difference in postoperative air-bone gap (ABG), sensorineural hearing loss (SNHL), or postoperative vertigo between procedures performed under local versus general anesthesia. No studies have evaluated or compared the cost-effectiveness of stapes surgery for otosclerosis performed under local versus general anesthesia.

This study hypotheses that patients undergoing stapes surgery under local anesthesia will have equivalent outcomes to those under general anesthesia, with the potential for reduced costs and operative time.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with otosclerosis and indicated for stapes surgery.
* Patients who underwent primary stapes surgery between January 1, 2022, and December 31, 2023.
* Surgery performed by utilizing the CO2 laser technique (Stapedotomy).
* Patients with complete medical records and audiometry data.
* Subjects do not object to the use of their personal data.

Exclusion Criteria:

* Patients with incomplete medical records (pre- or postoperative audiologic data were unavailable).
* Patients with other concurrent middle ear pathologies.
* Patients who underwent revision surgery for otosclerosis.
* performed by utilizing the microdrill technique or stapedectomy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent stapes surgery for otosclerosis from January 1, 2022, to December 31, 2023
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
To demonstrate the cost-effectiveness of performing stapes surgery for otosclerosis under local anesthesia. | From the first day of hospitalisation (date of entry) for stapes surgery until the last day of hospitalisation (date of discharge) on average, up to 2 days
  To compare the duration of hospital stay (in day) for patients undergoing the procedure under local anesthesia versus general anesthesia, and calculate the corresponding costs (in euros).
To analyse and describe the outcomes of stapes surgery for otosclerosis performed under both local and general anesthesia, and to compare these results with those reported in the literature. | From the first day of hospitalisation (date of entry) for stapes surgery until the last day of hospitalisation (date of discharge)on average, up to 2 days
  The percentage of air-bone gap closure postoperatively in both the local anesthesia and general anesthesia groups undergoing the procedure under local anesthesia versus general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Tavernier, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No